CLINICAL TRIAL: NCT02088944
Title: a Single-center Registered Clinical Research of Chinese Patients With Moderate to Severe Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: yimi-2
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Serological C Reactive Protein or Erythrocyte Sedimentation Rate
MeSH Terms: interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks

GROUPS / COHORTS (1):
- exposed to IFX
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab

SUMMARY:
Many studies reveal that infliximab (IFX, an immunoglobulin gamma-1 antibody)can response well to Crohn's Disease(CD) patients who are intolerant of corticosteroids and immunosuppressant,or steroids-dependent .More over,A complex fistula in CD is an indication for early IFX therapy in conjunction with surgical drainage.Some papers claim that IFX may prevent enterectomy CD patients from relapsing. Those with risk factors which at diagnosis associated with " disabling disease "include age < 40 years, initial need for steroid therapy, and the presence of perianal disease are recommended to use IFX early.

IFX is approved by State Food And Drug Administration(SFDA) in 2007 ,but the safety is still controversial by then.Some studies proclaim that the side effect may be infections,acute infusion reactions,anaphylactic reactions,autoimmunity,drug-induced lupus,congestive heart failure,abortion and demyelination,etc.

So some problems still need to be settled as follows:1)all the the infliximab dates are from other countries,there is rare date from the Chinese,especially the large quantity of random controlled studies and the CD patients with enterectomy.2)despite of the large number of databases from the international ,when to stop and the predictor of the response is still obscure.3)The high cost of IFX may hinder its applications,especially for the moderate to severe active CD patients who take mesalazine and/or immunosuppressant to maintain remission.In addition,the pathogenic age segments in the occurence of CD: from 15~ 50 years old ,so they suffer from the disability of self-improvements.

The main object of the clinical trial is to complete the database of Chinese CD patients ,especially the safety and efficacy of IFX and those with enterectomy.Then we can record the clinical manifestations of the moderate to severe CD patients with the use of IFX or conventional drugs,including the dose,course and Concomitant treatment.We can also study the predictor and the appropriate time to stop using IFX .We can make the mode of cost-benefit help the patients choose the best project.

ELIGIBILITY:
Inclusion Criteria:

* CD patients excluded from other diseases who are documented diagnosed with the tissue biopsy from colonoscopy or surgery,or those without tissue biopsy are followed over 6-12months finding that the clinical changs are in line with CD.
* The moderate to severe CD patients (Best Crohn's disease activity index>220）

Exclusion Criteria:

* Patients who are not willing to anticipate the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: moderate to severe CD patients
Sampling Method: Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
CD endoscopic index of severity(CDEIS)<4 | 4 years

SECONDARY OUTCOMES:
no endoscopic ulcer | 4 years